CLINICAL TRIAL: NCT04492436
Title: A Randomized, Double-blind, Placebo-controlled, Multi-national, Multi-center, Parallel-group, Phase 2b Assessing ART-123's Effect on Preventing Sensory Symptoms of OIPN in Unresectable mCRC Subjects Receiving Oxaliplatin-containing Chemo
Brief Title: A Trial Measuring ART-123 Ability to Prevent Sensory Neuropathy in Unresectable mCRC Subjects w/Oxaliplatin-based Chemo
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study design was changed
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2001B
Record Dates: First submitted 2020-07-22; First posted 2020-07-30 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — ART123

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Reconstituted lyophilized ART-123 with sterile water for injection administered by intravenous drip infusion over approximately 30 minutes on Day 1 of each chemotherapy cycle.
  Interventions: Drug: thrombomodulin alfa
- High Dose (Experimental): Reconstituted lyophilized ART-123 with sterile water for injection administered by intravenous drip infusion over approximately 30 minutes on Day 1 of each chemotherapy cycle.
  Interventions: Drug: thrombomodulin alfa
- Placebo (Placebo Comparator): Reconstituted lyophilized placebo with sterile water for injection administered by intravenous drip infusion over approximately 30 minutes on Day 1 of each chemotherapy cycle.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: thrombomodulin alfa — Weight based dose of reconstituted treatment administered through intravenous drip infusion on Day1 of each chemotherapy cycle
  Other Names: ART-123
  Arms: High Dose; Low Dose
Drug: Placebo — Weight based dose of reconstituted treatment administered through intravenous drip infusion on Day1 of each chemotherapy cycle
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of ART-123 on sensory symptoms of oxaliplatin-induced peripheral neuropathy (OIPN) in patients with unresectable metastatic colorectal cancer who receive oxaliplatin-containing chemotherapy

DETAILED DESCRIPTION:
To compare the efficacy and safety of ART-123 (low and high dose) to placebo on sensory symptoms of oxaliplatin-induced peripheral neuropathy (OIPN) in patients with unresectable metastatic colorectal cancer who receive oxaliplatin-containing chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Unresectable metastatic colorectal cancer; pathologically confirmed adenocarcinoma of the colon or rectum
* ECOG performance status of 0 or 1
* The most recent laboratory findings (including for liver and kidney) within 14 days prior to randomization remain within acceptable ranges
* Willingness of the patient and the sexual partner to use a highly effective contraceptive method during the course of the study
* Able to sufficiently understand the clinical study and give written informed consent

Exclusion Criteria:

* Prior treatment history with nerve toxic chemotherapeutic agent
* Peripheral neuropathy or central nervous system damage
* Psychiatric disorder
* History of major hemorrhage
* High risk of hemorrhage
* History of other malignancies
* Active ulcer
* Patients using anti-coagulants and fibrinolytic drugs
* Active Hepatitis B, or known HBs antigen positive
* Prior treatment history with thrombomodulin alfa
* Administration of another investigational medicinal product within 30 days prior to randomization
* Patient is pregnant (positive urine human chorionic gonadotropin) or breastfeeding or intends to get pregnant during the Treatment period
* Patients otherwise deemed as inappropriate to participate in the study by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
FACT/GOG-NTX-12 (4 items) Total Score at Cycle 9 | Cycle 9 (each cycle is 2 weeks)
  Change from baseline in total score of the first 4 items of the FACT/GOG-NTX-12 at the end of Cycle 9

SECONDARY OUTCOMES:
FACT/GOG-NTX-12 (4 items) Total Score at 9 Months | 9 months
  Change from baseline in total score of the first 4 items of the FACT/GOG-NTX-12 at 9 months
FACT/GOG-NTX-12 (4 items) Proportional Score at Cycle 9 (each cycle is 2 weeks) | Cycle 9 (each cycle is 2 weeks)
  Proportion of subjects scoring 3 or 4 in at least 1 of the first 4 items of the FACT/GOG-NTX-12 at the end of Cycle 9
FACT/GOG-NTX-12 (4 items) Cumulative Score at Cycle 9 | Cycle 9 (each cycle is 2 weeks)
  Cumulative incidence of scoring 3 or 4 in at least 1 of the first 4 items of the FACT/GOG-NTX-12 through Cycle 9
FACT/GOG-NTX-12 (12 items) Total Score at Cycle 9 | Cycle 9 (each cycle is 2 weeks)
  Change from baseline in total score of FACT/GOG-NTX-12 at the end of Cycle 9
NRS (Pain) Scores (feet) at Cycle 9 | Cycle 9 (each cycle is 2 weeks)
  Change from baseline score of NRS (Pain) in feet at the end of Cycle 9
NRS (Pain) Scores (hands) at Cycle 9 | Cycle 9 (each cycle is 2 weeks)
  Change from baseline score of NRS (Pain) in hands at the end of Cycle 9
Side Effect Questionnaire Score | Cycle 9 (each cycle is 2 weeks)
  Change from baseline score of Side effect questionnaire at the end of Cycle 9
CTCAE: Peripheral Sensory Neuropathy | Cycle 9 (each cycle is 2 weeks)
  Proportion of subjects with each Grade of CTCAE peripheral sensory neuropathy at the end of Cycle 9
CTCAE: Peripheral Motor Neuropathy | Cycle 9 (each cycle is 2 weeks)
  Proportion of subjects with each Grade of CTCAE peripheral motor neuropathy at the end of Cycle 9
mTCNS Score | Cycle 9 (each cycle is 2 weeks)
  Change from baseline in total score of mTCNS at the end of Cycle 9
Grooved Pegboard Change | Cycle 9 (each cycle is 2 weeks)
  Change from baseline score in the time to complete the Grooved Pegboard test with the non-dominant hand at the end of Cycle 9
EQ-5D-5L Change | Cycle 9 (each cycle is 2 weeks)
  Change from baseline in EQ-5D-5L index value at the end of Cycle 9

CONTACTS AND LOCATIONS:
Overall Officials: David Fineberg, MD, Study Director — Veloxis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No